CLINICAL TRIAL: NCT01315522
Title: Re-intervention for Occluded Biliary Metal Stent in Malignant Distal Bile Duct Obstruction: a Prospective Randomized Multi-center Trial Comparing Covered and Uncovered Metal Stent
Brief Title: Covered vs. Uncovered SEMS for Occluded Biliary Metal Stents
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ji Kon Ryu, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ERBD2SEMS
Record Dates: First submitted 2010-06-01; First posted 2011-03-15 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Biliary Tract Neoplasms; Jaundice, Obstructive
Keywords: Stents; Endoscopy; Cholangiopancreatography; Endoscopic Retrograde
MeSH Terms: conditions — Biliary Tract Neoplasms; Jaundice, Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ComVi stent (Active Comparator): ComVi stent (Niti-S stent, ComVi type, Taewoong Medical Inc, Korea)
  Interventions: Device: ComVi stent
- Uncovered SEMS (Active Comparator): uncovered nitinol metal stent (HANAROSTENT, M.I. Tech Co., Ltd., Korea)
  Interventions: Device: Uncovered SEMS

INTERVENTIONS:
Device: ComVi stent — Endoscopic insertion of ComVi stent
  Arms: ComVi stent
Device: Uncovered SEMS — Endoscopic insertion of uncovered SEMS
  Arms: Uncovered SEMS

SUMMARY:
Endoscopic retrograde biliary drainage (ERBD) is now widely accepted as the standard intervention for the relief of obstructive jaundice in patients with unresectable malignant biliary obstruction. Although plastic stents (PSs) were developed earlier, self-expandable metal stents (SEMSs) are now used widely as the initial choice for ERBD in this setting, as SEMSs offer longer patency.However, SEMSs do become occluded in some patients. There are a limited number of reports on the management of occluded SEMS with various results. The aim of this study is to compare the efficacy of ComVi stents SEMSs with uncovered SEMS in subsequent ERBD after the occlusion of initial SEMSs.

DETAILED DESCRIPTION:
Endoscopic placement of self-expandable metallic stents (SEMSs) is the mainstay of palliative measures for alleviating obstructive jaundice secondary to advanced cholangiocarcinoma. Previous meta-analysis showed no significant difference in stent patency between covered and uncovered SEMS, which are currently available. However, information on secondary SEMS insertion is still scarce, and there has been no prospective trial comparing efficacy of secondary stenting between covered and uncovered SEMS for the management of occluded metal stent in malignant biliary obstruction. Previously, only two small retrospective studies addressed this issue. Given the absence of prospective trial on re-intervention for occluded SEMS in malignant biliary obstruction, we aimed to prospectively compare the efficacies and complication rates of secondary ComVi stent (cSEMS) and uSEMS for the management of such condition.

ELIGIBILITY:
Inclusion Criteria:

* Patients with SEMS occlusion, which was inserted either endoscopically or percutaneously, for the relief of malignant nonhilar biliary obstruction
* Patients in whom the above SEMS had been inserted for no less than 7 days
* Patients with one of the following:

  1. cholangitis (as defined by fever, tenderness in the right upper quadrant or epigastrium, and/or a ≥ twofold increase in the serum bilirubin level above the baseline after initial SEMS insertion)
  2. a ≥ twofold increase in the serum bilirubin level above the baseline after initial SEMS insertion
* Patients in whom the cause of initial ERBD occlusion was identified, such as tumor overgrowth, ingrowth, and/or sludge
* Age ≥ 20 years

Exclusion Criteria:

* Unable to give informed consent
* Patients with sepsis and/or shock not responding to medical treatment or Eastern Cooperative Oncology Group (ECOG) Performance Status 4
* Patients with estimated survival < 4 weeks
* Patients who had undergone curative or palliative surgical intervention
* Hilar or perihilar biliary obstruction
* Patients who had undergone endoscopic nasobiliary drainage,plastic stent insertion, or percutaneous transhepatic biliary drainage prior to second SEMS insertion
* Covered SEMS as initial SEMS
* Migration or food impaction as the cause of initial SEMS occlusion

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2010-06; Primary Completion 2014-11 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
The stent patency | up to 53 months
  period between stent insertion and stent occlusion or death of the patient

SECONDARY OUTCOMES:
Technical success | for the duration of ERCP procedure, an expected average of 30 minutes
  Technical success was achieved when the SEMS was placed across the stricture with appropriate radiographic positioning and immediate biliary decompression
clinical success | within 2 weeks since initial ERBD
  Clinical success was achieved in the case of ≥ 50% reduction or normalization of total bilirubin level (≤ 1.2 mg/dL)
time-to-stent occlusion | up to 53 months
patient survival | up to 53 months
adverse events | within 4 weeks since initial ERBD
  stent migration, bleeding, pancreatitis, cholecystitis, or cholangitis

CONTACTS AND LOCATIONS:
Overall Officials: Ji Kon Ryu, MD, PhD, Principal Investigator — Seoul National University Hospital, Seoul National University College of Medicine
Locations (3):
- South Korea (3):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul

REFERENCES:
- [Derived] Lee BS, Ryu JK, Jang DK, Chung KH, Yoon WJ, Kim J, Woo SM, Lee SH, Lee WJ, Kim YT. Reintervention for occluded metal stent in malignant bile duct obstruction: A prospective randomized trial comparing covered and uncovered metal stent. J Gastroenterol Hepatol. 2016 Nov;31(11):1901-1907. doi: 10.1111/jgh.13392. PMID 27029890